CLINICAL TRIAL: NCT06751680
Title: Rhomboid Intercostal and Subserratus Plane Block Versus Paravertebral Block for Thoracic Herpes Zoster: a Randomized Comparative Trial
Brief Title: Rhomboid Intercostal and Subserratus Plane Block Versus Paravertebral Block for Thoracic Herpes Zoster
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaguang Duan (Other)
Responsible Party: Sponsor-Investigator, Xiaguang Duan, Deputy Chief of Anesthesiology, Inner Mongolia Baogang Hospital
Organization: Inner Mongolia Baogang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-MER-301
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-11

CONDITIONS: Thoracic Herpes Zoster
Keywords: Herpes Zoster; Paravertebral Block; Postherpetic Neuralgia; Regional Anesthesia; Rhomboid Intercostal and Subserratus Plane Block
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic

STUDY DESIGN:
Intervention Model Description: RISS group The RISS block is a composite nerve block technique that involves two injection sites, located in the inter-rhomboid plane and the sub-serratus plane, respectively. The choice of block plane depended on the patient's site of pain.
  PVB group Paravertebral Block
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- RISS group (Experimental): Rhomboid Intercostal and Subserratus Plane Block
  Interventions: Device: Rhomboid Intercostal and Subserratus Plane Block
- PVB group (Active Comparator): Paravertebral Block
  Interventions: Device: PVB block

INTERVENTIONS:
Device: Rhomboid Intercostal and Subserratus Plane Block — Upon entry, electrocardiogram (ECG), blood pressure, and oxygen saturation were monitored. The patient is placed in the prone position with their arms abducted and internally rotated. Ultrasound equipment (SonoSite Edge II; Fujifilm SonoSite, Bothell, WA, USA) with a linear 13-6 MHz transducer (HFL50x; Fujifilm SonoSite, Bothell, WA, USA) was used. Each nerve block was performed by initially injecting a 5 mL test dose, observing for clinical signs of pain relief in the affected thoracic dermatome, and then injecting the remaining volume of medication after confirmation of the injection site. Patients received ultrasound-guided nerve blocks every 48 hours, for a total of three treatments.The RISS block is a composite nerve block technique that involves two injection sites, located in the inter-rhomboid plane and the sub-serratus plane, respectively. The choice of block plane depended on the patient's site of pain.
  Arms: RISS group
Device: PVB block — The patient is placed in the prone position with their arms abducted and internally rotated. Ultrasound equipment (SonoSite Edge II; Fujifilm SonoSite, Bothell, WA, USA) with a linear 13-6 MHz transducer (HFL50x; Fujifilm SonoSite, Bothell, WA, USA) was used. Each nerve block was performed by initially injecting a 5 mL test dose, observing for clinical signs of pain relief in the affected thoracic dermatome, and then injecting the remaining volume of medication after confirmation of the injection site. Patients received ultrasound-guided nerve blocks every 48 hours, for a total of three treatments.After confirming needle tip placement, 10 mL of 0.5% ropivacaine with 10 mg of triamcinolone acetonide was slowly injected in divided doses, observing for the spread of the local anesthetic to ensure adequate distribution within the PVS for effective block. If multiple nerves were involved, the injection sites were spaced one thoracic vertebral segment apart.
  Arms: PVB group

SUMMARY:
Postherpetic neuralgia (PHN) is a common and debilitating complication of herpes zoster, characterized by persistent and severe pain. The rhomboid intercostal and subserratus plane (RISS) block, a novel ultrasound-guided regional anesthesia technique, has shown promise for various pain conditions, but its effectiveness for treating thoracic PHN remains relatively unexplored, and comparative studies against Paravertebral (PVB) block are lacking. This study aims to compare the efficacy and safety of RISS block versus PVB block for thoracic herpes zoster.

DETAILED DESCRIPTION:
This is a prospective, randomized, comparative, double-blinded (patient and clinician), superiority and non-inferiority clinical trial. This study compares the superiority and non-inferiority of RISS block versus PVB block for analgesia in the context of PHN. Patients were recruited from Baogang Hospital, Inner Mongolia. This study was approved by the Medical Ethics Committee of Baogang Hospital, Inner Mongolia (2023-MER-301) on December 19, 2023, and adhered to the Declaration of Helsinki and the Consolidated Standards of Reporting Trials (CONSORT) guidelines. All participants provided informed consent voluntarily.

Thirty patients with PHN, classified as ASA I-III, aged 44-82 years, and scheduled to receive either a RISS block or a PVB block between January 2024 and November 2024, were selected, with 15 patients per group. Inclusion criteria: Patients with typical manifestations of herpes zoster (HZ) , such as vesicular and painful rash; herpes zoster neuralgia lasting more than one month and unresponsive to conventional treatment; a VAS score ≥ 4; and thoracic nerve root involvement. Exclusion criteria: Patients who refused to provide written informed consent; were unable to cooperate with assessments; had a history of systemic autoimmune disease, organ transplantation, or cancer; had received other invasive treatments (e.g., spinal cord stimulation); had a central nervous system disorder; had coagulopathy; had a skin infection at the puncture site; or were pregnant/lactating.

Patients with PHN refractory to pharmacological treatment were considered for either RISS block or PVB block. All patients received famciclovir and gabapentin. Patients received standard antiviral treatment with famciclovir 500 mg three times daily for 7 days. Gabapentin was initiated at a dose of 300 mg/day, typically divided into three administrations. The dose was gradually increased to a maximum of 1800 mg/day as needed and tolerated. All procedures were performed in an outpatient operating room, and all participating physicians had undergone standardized training. Upon entry, electrocardiogram (ECG), blood pressure, and oxygen saturation were monitored. The patient is placed in the prone position with their arms abducted and internally rotated. Ultrasound equipment (SonoSite Edge II; Fujifilm SonoSite, Bothell, WA, USA) with a linear 13-6 MHz transducer (HFL50x; Fujifilm SonoSite, Bothell, WA, USA) was used. Each nerve block was performed by initially injecting a 5 mL test dose, observing for clinical signs of pain relief in the affected thoracic dermatome, and then injecting the remaining volume of medication after confirmation of the injection site. Patients received ultrasound-guided nerve blocks every 48 hours, for a total of three treatments.

Follow-up assessments were conducted at the pain clinic by two specially trained nurses who were blinded to patient allocation, at baseline (before therapy), on the day of treatment (Day 1), and at 7 days (Day 7), 30 days (Day 30), and 90 days (Day 90) post-treatment, either in person or via telephone.

Primary outcomes

ELIGIBILITY:
Inclusion Criteria:

* Patients with typical manifestations of herpes zoster (HZ), such as vesicular and painful rash
* herpes zoster neuralgia lasting more than one month and unresponsive to conventional treatment
* a VAS score ≥ 4
* thoracic nerve root involvement

Exclusion Criteria:

* refused to provide written informed consent
* unable to cooperate with assessments
* history of systemic autoimmune disease, organ transplantation, or cancer
* received other invasive treatments (e.g., spinal cord stimulation)
* central nervous system disorder
* coagulopathy
* skin infection at the puncture site
* pregnant/lactating

Ages: 44 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale(NRS) | At baseline (before therapy), on the day of treatment, at 7 days post-treatment, 30 days post-treatment, and 90 days post-treatment
  The NRS, Numerical Rating Scale, is a rating system from 0 to 10, where 0 represents "no pain" and 10 represents the worst possible pain.

SECONDARY OUTCOMES:
The Zoster Brief Pain Inventory (ZBPI) | At baseline (before therapy), on the day of treatment, at 7 days post-treatment, 30 days post-treatment, and 90 days post-treatment
  The daily activity questionnaire included seven items: general activity, mood, walking ability, normal work, relationships with others, sleep, and enjoyment of life. Each question concerning daily activity was scored on a scale from 0 to 10, where 0 indicated no interference and 10 indicated complete interference.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangyu Wang, Undergraduate, Principal Investigator — Inner Mongolia Baogang Hospital
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: January 2025-January 2027
Access Criteria: A proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed.